CLINICAL TRIAL: NCT06949306
Title: Intervention of a Digital Health Management Program in Patients With Cardiometabolic Disorders: a Real-world Study
Brief Title: Intervention Study on Digital Health Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, professor of Medicine, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSS_3.0
Record Dates: First submitted 2025-04-13; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-03

CONDITIONS: Hypertension; Hyperlipidemia
Keywords: Cardiometabolic abnormalities; Digital Interventions
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Dental Assistants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardiovascular digital management group (Experimental): Participants used a bracelet and an APP assistant for lifestyle interventions
  Interventions: Other: Bracelet, assistant, APP: the "golden triangle" of smart life

INTERVENTIONS:
Other: Bracelet, assistant, APP: the "golden triangle" of smart life — The lifestyle intervention was carried out through the bracelet, Little Assistant and Keyhealth APP for 24 weeks, and the daily data synchronization of the APP and weekly AI feedback were performed. After 24 weeks, blood glucose, blood lipid, blood pressure, CAI and other indicators were monitored.

SUMMARY:
The aim of this study is to construct a digital precision intervention system for cardiometabolism disorders based on the characteristics of the Chinese population, focusing on the core components of metabolic syndrome such as hypertension, hyperglycemia, and obesity. Through dynamic monitoring of wearable devices, the individualized risk factors (including genetic predisposition, lifestyle, and psychological factors) of metabolic disorders were systematically analyzed, and dynamic intervention strategies were formulated accordingly. The closed-loop management of "monitor-feedback-optimization" based on the digital platform will provide patients with one-stop metabolic risk assessment and panoramic health management plan, realizing a paradigm shift from "generalized intervention" to "precise regulation". By reducing the abnormal fluctuations of key metabolic indicators such as blood pressure, blood glucose, and blood lipids, the risk of cardiovascular events will eventually be reduced, the long-term quality of life of patients will be improved, and a practical path of "digital therapy" can be promoted for the prevention and control of chronic diseases in China

ELIGIBILITY:
Inclusion Criteria:1. Age 18-65 years old; 2. Meet one of the following three conditions:

1. Diastolic hypertension (systolic blood pressure < 140 MMHG and diastolic blood pressure ≥90mmHg)
2. Glycosylated hemoglobin (6.0-6.5)
3. Obesity (BMI≥28kg/m²)
4. Mild hyperlipemia: total cholesterol (TC) ≥5.2 mmol/L and < 6.2 mmol/L, or low-density lipoprotein cholesterol (LDL-C) ≥3.4 mmol/L and < 4.1 mmol/L 3. Antihypertensive or lipid-lowering medications have not been started 4. Use a smartphone and volunteer

Exclusion Criteria:

1. Complicated with chronic liver and kidney disease, coronary heart disease, heart failure and severe valvular disease
2. Previous cardiovascular and cerebrovascular events
3. Diastolic blood pressure ≥99mmHg
4. Glycated hemoglobin ≥6.5
5. Other life expectancy such as cancer is less than 5 years
6. Participate in other clinical trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in diastolic blood pressure after 24 weeks | 24 weeks following intervention

SECONDARY OUTCOMES:
Values for changes in Hba1c or BMI or CAI after 24 weeks | 24 weeks following intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology,Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided